CLINICAL TRIAL: NCT03383523
Title: Phase1,Randomized,Open-Label,Parallel-Group,Relative Bioavailability Study to Investigate PK,Including Food Effect,Safety and Tolerability of Single Doses of New Immediate Release Tablet Formulations of Emodepside (BAY 44-4400),Compared to Oral Solution,in Healthy Male Subjects
Brief Title: Relative Bioavailability Study of Emodepside IR-tablets and Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Bayer (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDI-EMO-03; 2017-003091-31 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2017-12-26 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Filariasis
MeSH Terms: conditions — Filariasis | interventions — emodepside; Bay 44-4400; Praziquantel; toltrazuril

STUDY DESIGN:
Intervention Model Description: This is a single-centre, open-label, randomized, parallel-group relative bioavailability study in healthy men. The study will be done in 2 parts, as follows:
  Part 1 - single oral doses of 5 mg emodepside will be tested:
  * Part 1a - the LSF (reference formulation) and 2 new IR-tablet formulations (test formulations) will be administered in the fasted state.
  * Part 1b - the 2 new IR-tablet formulations will be administered in the fed state (high-fat, high-calorie meal).
  Part 2 - single oral doses of 10 mg emodepside will be tested: depending on the results from Part 1, one or both IR-tablet formulations will be administered in the fasted state.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1a - treatment A (Experimental): 5 mg emodepside LSF, fasted
  Interventions: Drug: Emodepside (BAY 44-4400)
- Part 1a - treatment B (Experimental): 5 mg emodepside IR-tablet #406, fasted
  Interventions: Drug: Emodepside (BAY 44-4400)
- Part 1a - treatment C (Experimental): 5 mg emodepside IR-tablet #416, fasted
  Interventions: Drug: Emodepside (BAY 44-4400)
- Part 1b - treatment D (Experimental): 5 mg emodepside IR-tablet #406, fed
  Interventions: Drug: Emodepside (BAY 44-4400)
- Part 1b - treatment E (Experimental): 5 mg emodepside IR-tablet #416, fed
  Interventions: Drug: Emodepside (BAY 44-4400)
- Part 2 - treatment F (Experimental): 2 x 5 mg emodepside IR-tablet #406, fasted (may be tested or not, depending on the results of the part 1)
  Interventions: Drug: Emodepside (BAY 44-4400)
- Part 2 - treatment G (Experimental): 2 x 5 mg emodepside IR-tablet #416, fasted (may be tested or not, depending on the results of the part 1)
  Interventions: Drug: Emodepside (BAY 44-4400)

INTERVENTIONS:
Drug: Emodepside (BAY 44-4400) — 2 tablets compared to the liquid formulation
  Other Names: Profender® (in combination with praziquantel) FOR VETERINARY USE; Procox® (in combination with toltrazuril) FOR VETERINARY USE

SUMMARY:
This study evaluates 2 new immediate release (IR)-tablet formulations of emodepside and they will be compared to the oral liquid service formulation (LSF) used in the FIH Single Ascending Dose study (DNDi-EMO-001 study) (CT.gov identifier: NCT02661178)

DETAILED DESCRIPTION:
There is an urgent need for a macrofilaricidal drug, killing or sterilizing permanently O. volvulus adult worms, which could be used in individual case management and, after appropriate testing, as an alternative drug to ivermectin in MDA programs. Emodepside is a promising candidate to kill the adult and sexually mature O. volvulus. Emodepside was shown to be macrofilaricidal against a variety of filarial nematodes and is a registered drug for animal health, commercialized by Bayer AG under the name of Profender® (in combination with praziquantel) or Procox® (in combination with toltrazuril).

A first-in-human (FIH) double-blind, placebo-controlled study of single ascending doses of emodepside in healthy Caucasian men has been conducted and the preliminary results are favourable, and support continuing the Phase I development program. For this reason, new tablet formulations have been developped and the present study will evaluate bioavailability, PK safety and tolerability, and as well food effect of single doses of 2 new immediate release (IR)-tablet formulations of emodepside compared to the oral liquid service formulation (LSF) used in the FIH study.

ELIGIBILITY:
Inclusion Criteria:

1. Male, Caucasian volunteers, deemed healthy based on a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine.
2. 18 to 45 years of age
3. Normal body weight (Body Mass Index (BMI); Quetelet index) in the range 18.0 to 30.1 kg/m2 at screening
4. Mean blood pressure and heart rate (from the triplicate readings) in the supine position at the screening assessment outside one (or more) of the ranges: 90-140 mm Hg systolic BP 60-90 mm Hg diastolic BP 45-100 beats/min HR
5. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire trial
6. Willingness to give written consent to participate, after reading the information and consent form, and after having the opportunity to discuss the trial with the Investigator or his delegate
7. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS)
8. Willingness to follow contraception requirements of the study, from the first dose of the IMP until 90 days after dosing and inform HMR as soon as possible if their partner becomes pregnant in the 90 days after dosing

   Exclusion Criteria:
9. Administration of a licensed or unlicensed medicinal product as part of another clinical trial in the 3 months before the first dose of study medication, or within 5 half-lives of administration of a medicinal product given in the previous study (whichever is longer), or otherwise in the follow-up period for any clinical trial
10. Clinically relevant abnormal medical history, concurrent medical condition, acute or chronic illness, or history of chronic illness (such as diabetes mellitus or other abnormalities of glucose homeostasis) sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous
11. Past surgery (e.g. stomach bypass) or medical condition that might affect absorption of the study drug when taken orally
12. Presence of abnormal physical findings, ECG, or laboratory values at the screening assessment that could interfere with the objectives of the trial or the safety of the subject
13. Loss of more than 400 mL of blood within the 3 months before admission
14. Clinically relevant history of vital organ disease, or other organ or central nervous system disease (e.g. diabetes mellitus, liver disease, seizures, etc.)
15. Current or previous medical or psychiatric disorder that, in the opinion of the Investigator or the Sponsor, would increase the risk and ability to participate in and/or complete the study
16. Positive test for hepatitis B, hepatitis C or HIV
17. Febrile illness (e.g. fever) within 1 week before the first dose of study medication
18. History of a severe allergy, non-allergic drug reaction, severe adverse reaction to any drug, or multiple drug allergies
19. Hypersensitivity to any ingredient of the study medication, including the active ingredient (emodepside)
20. Presence or history of drug or alcohol abuse in the last year, or intake of more than 21 units (1 unit = 1/2 pint of beer, 1 small glass of wine or 1 measure of spirits) of alcohol weekly
21. Regular daily consumption of more than one litre of beverages containing xanthine
22. Daily consumption of more than 10 cigarettes or more than 6 grams (1/4 ounce) of tobacco
23. Use of a prescription medicine during the 28 days before the dose of study medication, or use of an over-the-counter medicine (with exception of acetaminophen (paracetamol)), during the 7 days before the dose of study medication
24. Use, within 14 days before the dose of study medication, of dietary supplements or herbal remedies (such as St John's Wort) that are known to be inducers or inhibitors of CYP3A4, or other co-medications known to be relevant substrates of CYP3A4 (see list in the Study Procedures Manual)
25. Use, within 14 days before the dose of study medication, of dietary supplements or herbal remedies that are known to be strong inhibitors of P-gp, or other co-medications known to be relevant substrates of P-gp (see list in the Study Procedures Manual)
26. Relevant pathological abnormalities in the ECG at screening, such as:

    second or third-degree atrioventricular (AV) block prolongation of the QRS complex > 120 msec, QTc-interval (QTcB or QTcF) > 450 msec. The mean of the triplicate ECG readings will be used to assess eligibility.
27. Evidence of drug abuse (via urine testing) at the screening assessment or admission to the ward
28. Use of excluded therapies that may impact on the interpretation of study results in the opinion of the Investigator or Sponsor
29. Objection by General Practitioner (GP) to subject entering trial
30. History of residing for 6 or more continuous months during the last 3 years in regions with endemic parasitic infections, as determined by the Investigator
31. Possibility that subject will not cooperate with the requirements of the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male only
Enrollment: 77 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Dennison, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research (HMR) Limited, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential volunteers contacted HMR by telephone or email if they were interested in the study. HMR contacted eligible volunteers who had registered an interest in doing this study to invite them to take part. Recruitment of participants started on 26 October 2017 (FSFV) and finished on 26 March 2018 (LSLV).
Pre-assignment Details: screening details: to check they were healthy and eligible for the study, volunteers had a full examination at screening including physical and neurological examination, vital signs, 12-lead ECG monitoring, safety blood tests (hematology, biochemistry, coagulation and urinalysis), drug screen, alcohol breath test and serology
Period: Overall Study
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Started | 11 | 11 | 10 | 12 | 11 | 12 | 10
Completed | 10 | 11 | 9 | 12 | 11 | 12 | 10
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy Caucasian males subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G | Total
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 10 | 12 | 11 | 12 | 10 | 77
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [21 to 38] | 32.4 [18 to 44] | 32.2 [23 to 43] | 32.6 [23 to 44] | 30.5 [18 to 42] | 30.5 [20 to 44] | 29.8 [18 to 38] | 31.1 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 11 | 11 | 10 | 12 | 11 | 12 | 10 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 10 | 12 | 11 | 12 | 10 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 11 | 11 | 10 | 12 | 11 | 12 | 10 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 11 | 10 | 12 | 11 | 12 | 10 | 77

OUTCOME MEASURES:

1. Primary Outcome: PK (AUC0-7d) of Two New Tablet Formulations of Emodepside in Comparison to the Liquid Formulation (LSF) Oral Solution.
Description: Means AUC from zero to 7 days (AUC0-7d) = means area under the plasma concentration-time curve from time zero (pre-dose) to 7 days. To create the curve, the following PK Timepoints have been collected: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3,4,6,8,12,36,48,72,120 and 168h post dose
Time Frame: means from zero to 7 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/ml
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
h.ng/ml | 1215 (37.2) | 852 (19.1) | 931 (23.3) | 674 (32.1) | 733 (34.9) | 1609 (35.9) | 1943 (26.5)

2. Primary Outcome: PK (Cmax) of Two New Tablet Formulations of Emodepside in Comparison to the Liquid Formulation (LSF) Oral Solution.
Description: Cmax means maximum observed plasma concentration. To create the PK curve, the following PK timepoints have been collected: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3,4,6,8,12,36,48,72,120 and 168h post dose
Time Frame: 7 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
ng/ml | 88.5 (20.1) | 41.9 (20.0) | 54.2 (35.3) | 27.1 (26.8) | 36.2 (39.8) | 71.7 (28.5) | 135 (35.3)

3. Secondary Outcome: Safety and Tolerability as Measured by Number of Participants With Treatment-related Adverse Events
Description: number of participants with treatment-related adverse events
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
Participants | 0 | 3 | 1 | 0 | 1 | 0 | 1

4. Secondary Outcome: Safety and Tolerability as Measured by Number of Participants With Physical Examination Findings
Description: number of participants with abnormal physical examination (PE) findings. Standard examination done on head, ears, eyes, nose, thyroid, lymph node, back, neck, lungs, skin, abdomen, chest. The details are listed in protocol section 8.11.3
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
participants
  number of subject with abnormal PE findings | 0 | 0 | 1 | 0 | 1 | 0 | 0
  number subject with clinically significant finding | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Safety and Tolerability as Measured by Number of Participants With Neurological Examination Findings
Description: Number of participants with abnormal neurological examination (NE) findings
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
participants
  number of subject with abnormal NE findings | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number subject with clinically significant finding | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Safety and Tolerability as Measured by Number of Participants With Vital Signs Findings
Description: number of participants with vital signs (VS) findings. The vital signs ranges are the following Supine Systolic BP : 85-160mm HG, Supine Diastolic BP: 40-90mm HG, Supine HR: 35-100 beats/min. Details are described in the protocol section 8.11.2
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
participants
  number of subject with VS findings | 0 | 1 | 2 | 2 | 3 | 0 | 0
  number subject with clinically significant finding | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Safety and Tolerability as Measured by Number of Participants With 12-lead ECG Findings
Description: number of participants with 12-lead ECG findings. The ECG reference ranges used are the following: ventricular rate: 45-100beats/min, PR interval:120-220msec, QRS:<120msec, QTc:<430msec
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
participants
  number of subject with abnormal ECG findings | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number subject with clinically significant finding | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Safety and Tolerability as Measured by Number of Participants With Clinical Laboratory Tests Findings
Description: number of participants with relevant abnormal laboratory tests results
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 11 | 12 | 10
participants
  number of subject with abnormal lab values | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number subject with clinically significant finding | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were reported from screening (up to 28 days before dosing) up to Follow up visit (7 days after dosing)
Arm/Group | Part 1a - Treatment A | Part 1a - Treatment B | Part 1a - Treatment C | Part 1b - Treatment D | Part 1b - Treatment E | Part 2 - Treatment F | Part 2 - Treatment G
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/12 | 0/11 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/12 | 0/11 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 3/11 | 5/11 | 2/10 | 1/12 | 5/11 | 0/12 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a - Treatment A (N=11) | Part 1a - Treatment B (N=11) | Part 1a - Treatment C (N=10) | Part 1b - Treatment D (N=12) | Part 1b - Treatment E (N=11) | Part 2 - Treatment F (N=12) | Part 2 - Treatment G (N=10)
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 2
diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0
visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
catheter site (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
abdominal disconfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
feeling of relaxation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the PI and the sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03383523/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03383523/SAP_001.pdf